CLINICAL TRIAL: NCT04909034
Title: A Randomized, Placebo Controlled Study to Evaluate the Safety and Potential Efficacy of MS-20 in Combination with Pembrolizumab for the Treatment of Non-Small-Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB103CLAS08
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: NSCLC Stage IIIB~IV
Keywords: NSCLC; MS-20; Add-on; pembrolizumab; metastatic; microbiome; microbiota
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MS-20 oral solution (Experimental): Oral Solution 4 c.c, divided twice daily (BID) for 48 weeks.
  Interventions: Drug: MS-20
- Placebo (Placebo Comparator): Oral Solution 4 c.c, divided twice daily (BID) for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MS-20 — Fermented soybean extract MicrSoy-20(MS-20), which uses a variety of lactic acid bacteria and yeasts to metabolize organic soybeans
  Other Names: Chemo young
  Arms: MS-20 oral solution
Drug: Placebo — Oral solution without active ingredients
  Arms: Placebo

SUMMARY:
MS-20 was approved as the first oral cancer adjuvant new drug indicated for ameliorating fatigue and appetite loss associated with cancer chemotherapy via reshaping human gut ecosystem and restoring immunity. MS-20 has also been shown to be anti-PD-1 booster by activating tumor-infiltrating lymphocytes (TILs) in mice cancer models, particularly promoting migration of TILs into tumors and increasing the amount of TILs inside tumors. Therefore, this study is designed to explore the potential clinical outcomes, safety and relationship between gut microbiome in NSCLC patients under combination therapy with pembrolizumab and MS-20.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are over 20 years old (inclusive) at the time of signing the informed consent form.
2. The subject is diagnosed pathologically or cytologically with non-small cell lung cancer (NSCLC).
3. According to the 8th edition of the American Joint Committee on Cancer [AJCC], staging is metastatic III.B-IV NSCLC that cannot be surgically removed.
4. The subject with metastatic non-squamous carcinoma whose EGFR/ALK/ROS 1 tumor gene is the original type, or subject with squamous cell carcinoma whose EGFR/ALK tumor gene is the original type.
5. At least one measurable lesion per RECIST v 1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. The subject whose biomarker performance: The PD L1 performance detected by Dako 22C3 or Ventana SP263 and other third-level in vitro diagnostic medical devices (class III) must meet tumor proportion scores (TPS) ≥ 50%.
8. The life expectancy is not less than 3 months.
9. The subject whose liver and kidney functions must meet all of the following conditions:

   * Liver function: aspartate aminotransferase (AST) value < 2.5 x ULN, alanine aminotransferase (ALT) value < 2.5 x ULN and total bilirubin (T-bilirubin) value < 1.5 x ULN. For the subjects who have liver metastases, total bilirubin value should be < 5 x ULN.
   * Kidney function: Serum creatinine value < 1.5 ULN. If subject's serum creatinine value is ≥ 1.5 x ULN, his/her creatinine clearance value should be > 40 mL/min based on Cockcroft and Gault formula.
10. Subject, if female of child-bearing potential, must agree to avoid sexual intercourse or be willing to use 2 medically accepted methods of contraception (e.g., Intra-uterine device or contraceptives) during the study. 【The definition of infertile：(1) Being menopause for more than 1 year；(2) Surgery for permanent contraception (e.g., abdominal tubal sterilization, bilateral Salpingooophorectomy, and tubectomy)；(3) Congenital structural abnormalities.】
11. Subject, if male, agrees not to donate sperm, be willing to avoid sexual intercourse or use appropriate contraception method (e.g., using condom) during the study treatment period.
12. Subject is active and capable to communicate with site staff, willing to be in compliance with the following two items based on investigator's judgment.

    1. To complete return visits and study examination per the study protocol.
    2. To collect stool specimens at home, refrigerate and deliver the sample.

Exclusion Criteria:

1. Presence of any symptomatic central nervous system metastasis or leptomeningeal metastasis.
2. Presence of any other malignant tumor. Unless the subject had completed radical treatment without any disease recurrence for at least 3 years. (Those who have successfully undergone radical resection or have received possible curative treatments for basal cell carcinoma, superficial bladder cancer, squamous-cell carcinoma, cervical intraepithelial neoplasia or other carcinoma in situ are not limited)
3. Presence of any autoimmune disease which requires systemic treatment within the past 2 years. Hormone replacement therapy (for example, insulin or physiological replacement of corticosteroid due to adrenal or pituitary disorders… etc.) is allowed and not considered as systemic treatment.
4. Have had any transplantation of allogeneic cell, tissue or solid organ.
5. History of known human immunodeficiency virus (HIV) infection.
6. Hepatitis B surface antigen (HBsAg) is positive or hepatitis B virus (HBV) DNA viral load is ≥ 500 IU/mL.Or Hepatitis C virus (HCV) antibody is positive and hepatitis C virus (HCV) ribonucleic acid (RNA) is also positive.
7. Subject has non-infectious pneumonia history which requires systemic steroids. Subject who currently have interstitial pneumonia or interstitial pneumonitis can join this study if investigator confirms subject's clinical condition is stable.
8. Presence of any severe cardiac dysfunction, Class III-IV of chronic heart failure based on New York Heart Association (NYHA) Functional Classification, which includes symptomatic coronary artery disease and severe ventricular arrhythmia; Presence of any myocardial infarction, unstable or poorly controlled angina within 6 months before subject screening visit (V0).
9. Have any gastrointestinal history or surgery which investigator believes may affect the absorption of the oral investigational product.
10. Enterocutaneous or non- enterocutaneous fistula which is defined as Grade 3 or above based on Common Terminology Criteria for Adverse Events (CTCAE, also known as Common Toxicity Criteria).
11. Currently presence of inflammatory bowel disease or gastric ulcer.
12. Have not yet recovered from major surgery or complications before subject screening visit(V0).
13. History of active tuberculosis (TB, Mycobacterium tuberculosis).
14. Presence of any mental disease or drug abuse disorder which may interfere with subject's ability for being compliant with study requirements.
15. Active infection which requires systemic treatment.
16. Allergies to soy products, severe allergies to antibody therapy, or known allergies or intolerances to any component of pembrolizumab.
17. Have received any biologic therapy within 3 weeks prior to the first dose of trial therapy.
18. Have received anti-PD-1, anti-PD-L1, or anti-PD-L2 drug therapy within 3 years before the screening visit (V0) or act on another drug treatment that stimulates signals or synergistically inhibits T cell receptors (e.g. CTLA-4 , OX 40, CD137).
19. Received radiotherapy within the 14 days before receiving the investigational drug, or received pulmonary radiotherapy> 30 Gy within 6 months before receiving the investigational drug (the subject must recover from all radiation-related toxicities to grade 1 or below, without corticosteroid therapy and radiation pneumonia has never occurred).
20. Diagnosed with immunodeficiency or are receiving any form of immunosuppressive therapy, systemic steroids (allowed to use up to 10 mg Prednisone or equivalent steroids per day) within 7 days before receiving the investigational drug.
21. Those who have received live-virus vaccines within 30 days before receiving the investigational drug or are expected to receive live-virus vaccines during the study period.
22. Have used antibacterial drugs including antibiotics and synthetic drugs (such as sulfonamides, quinolones), antifungal or antiviral drugs (not including topical medication) within the 14 days before receiving the investigational drug.
23. Use probiotics and probiotic-related products within 14 days before receiving this test drug (e.g. yogurt, yogurt, Yakult, probiotic fermented beverages, Wakamoto tablets, Shin Biofermin S tablets, inulin, oligosaccharide products).
24. Have used laxatives (such as MgO, Bisacodyl, Sennoside, Lactulose) within the 14 days before receiving the investigational drug.
25. Those who have had gastrointestinal infection and diarrhea within the 14 days before receiving the investigational drug (soft or watery stools more than three times within 24 hours).
26. Women who are pregnant, breastfeeding or expect to breastfeed during the study period.
27. Currently participating in clinical trials of other investigational product treatments, medical devices, health foods, or cosmetics.
28. Subjects who judged by the investigator to be unsuitable to participate in the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the objective response rate (ORR) in subjects with metastatic non-small cell lung cancer (NSCLC) treated with MS-20 combined with pembrolizumab. | 48 weeks
  According to RECIST 1.1, the objective response rate (ORR) assessed by contrast is defined as the proportion of patients whose tumors shrink to a predetermined amount and remain for a period of time, which is the sum of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression free survival (PFS) | 48 weeks
  According to Solid Tumor Efficacy Evaluation Criteria Version 1.1 (RECIST 1.1), is defined as the time from the beginning of the treatment period to the first documented progressive disease (PD) or death from any other non-PD cause (whichever occurs first).
Disease control rate (DCR) | 48 weeks
  According to the Solid Tumor Efficacy Evaluation Criteria Version 1.1 (RECIST 1.1), defined as the proportion of subjects whose optimal overall response was determined to be a complete response (CR), partial response (PR), or disease stabilization (SD).
Duration of response (DOR) | 48 weeks
  Assessed according to the Solid Tumor Efficacy Evaluation Criteria Version 1.1 (RECIST 1.1), defined as the minimum time from the first observation of a complete response (CR) or partial response (PR) to disease progression (PD) or death for subjects whose best overall response after treatment is complete response (CR) or partial response (PR). Otherwise, DOR will be the time of the last tumor evaluation.
Safety assessment- incidence of adverse events (TEAEs) | 48 weeks
  Following treatment with the investigational product. According to "The NCI Common Terminology Criteria for Adverse Events Fifth Edition Evaluation Form; Common Terminology Criteria for Adverse Events (CTCAE) V5.0" as a clinical evaluation tool.

OTHER OUTCOMES:
To evaluate the effect on the gut microbiota in subjects with metastatic non-small cell lung cancer treated with MS-20 combined with pembrolizumab. | 48 weeks
  To evaluate the effect on the gut microbiota in subjects with metastatic non-small cell lung cancer treated with MS-20 combined with pembrolizumab.
Safety | 48 weeks
  Safety will be assessed by physical examinations, laboratory tests, monitoring AEs, vital signs, and concomitant medication usage.

CONTACTS AND LOCATIONS:
Locations (7):
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Ministry of Health and Welfare Shuang-Ho Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No